CLINICAL TRIAL: NCT07195266
Title: A Naturalistic Study of Psychological Outcomes in Adult Outpatients Receiving Strategic Psychotherapy in Private Practice (POST)
Brief Title: Psychological Outcomes of Strategic Therapy in Adult Outpatients (POST Trial)
Acronym: POST
Status: Recruiting | Type: Observational
Sponsor: Società Scientifica di Psicoterapia Strategica (Other)
Responsible Party: Principal Investigator, Fabio Leonardi, Professor, Società Scientifica di Psicoterapia Strategica
Other Study IDs: POST 01
Record Dates: First submitted 2025-09-09; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Mental Disorder
Keywords: Strategic Therapy; Psychotherapy; Mental disorders
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Strategic Psychotherapy: patients receiving strategic psychotherapy in private practice settings
  Interventions: Behavioral: Strategic Psychoterapy

INTERVENTIONS:
Behavioral: Strategic Psychoterapy — Strategic psychotherapy as described in scientific literature

SUMMARY:
This observational study investigates the outcomes of Strategic Psychotherapy, a form of brief psychological treatment focused on specific goals for change, co-constructed with patients. The aim is to evaluate whether patients who receive this therapy in private practice settings experience improvements in their psychological well-being, symptoms, and daily functioning.

The study population includes all adult patients (≥18 years) who spontaneously seek treatment from two strategic therapists between January 2021 and December 2025. Eligible participants must present with psychological problems that meet the criteria for a clinical diagnosis.

Participants will complete two psychological questionnaires (SCL-90R and CORE-OM) before starting therapy and again at the end of their treatment.

Additional information will be collected, such as use of medication, the patient's own evaluation of the therapy, number of sessions attended, initial diagnosis, involvement of family members, and types of prescriptions used.

All data will be treated confidentially and used solely for research purposes.

DETAILED DESCRIPTION:
Strategic Psychotherapy is a form of brief, goal-oriented psychological treatment that emphasizes the collaborative construction of specific therapeutic goals and the implementation of targeted interventions to promote change. Despite its widespread clinical application, there is limited systematic evidence on patient outcomes in naturalistic private practice settings.

This observational study aims to contribute to the evidence base by examining the effectiveness of Strategic Psychotherapy in improving psychological well-being, reducing symptom distress, and enhancing everyday functioning. The study includes all adult patients (≥18 years) who independently seek treatment from two certified strategic therapists between January 2021 and December 2025. Inclusion is based on the presence of clinically relevant psychological problems consistent with a formal diagnosis.

Participants will be assessed at baseline and post-treatment using two standardized and validated outcome measures: the Symptom Checklist-90 Revised (SCL-90R) and the Clinical Outcomes in Routine Evaluation - Outcome Measure (CORE-OM). Additional clinical and process variables will be recorded, including initial diagnosis, medication use, number of sessions attended, involvement of family members, type of prescriptions, and patient's subjective evaluation of therapy.

Therapists will not manipulate or control the number of sessions or content of therapy beyond their usual clinical practice, thereby preserving the ecological validity of the study. The design is naturalistic and observational, without randomization or control groups. All data will be anonymized and handled in accordance with confidentiality and data protection standards. Findings are expected to provide insight into the real-world outcomes of Strategic Psychotherapy and contribute to the development of evidence-based practice guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older.
* Individuals voluntarily seeking psychological treatment in private practice with one of the participating strategic therapists.
* Presence of clinically relevant psychological problems consistent with a formal diagnosis (e.g., anxiety disorders, depressive disorders, stress-related conditions, relational difficulties).
* Ability to provide informed consent.

Exclusion Criteria:

* Individuals younger than 18 years.
* Patients with severe psychiatric conditions requiring immediate specialized care (e.g., acute psychosis, severe suicidal risk, substance dependence requiring detoxification).
* Patients currently enrolled in another clinical trial.
* Inability or unwillingness to complete the required questionnaires (SCL-90-R and CORE-OM).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will consist of adult patients (≥18 years) who voluntarily seek psychological treatment in private practice with two licensed strategic therapists in Livorno and Empoli, Italy. Participants are individuals presenting with clinically relevant psychological problems consistent with a formal diagnosis (e.g., anxiety, depression, stress-related or relational difficulties). Patients are not recruited through advertising or referral; they are self-referred clients seeking therapy during the period January 2021 to December 2025.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
1. Symptom Checklist-90-Revised (SCL-90-R) 2. Clinical Outcomes in Routine Evaluation - Outcome Measure (CORE-OM) | Baseline (prior to first psychotherapy session) and at end of treatment (average of 12-16 weeks, depending on number of sessions).
  1. Symptom Checklist-90-Revised (SCL-90-R) Description: A 90-item self-report scale assessing psychological symptoms across multiple domains. Each item is rated on a 5-point Likert scale (0 = "not at all" to 4 = "extremely"). Higher scores indicate greater symptom severity.
  2. Clinical Outcomes in Routine Evaluation - Outcome Measure (CORE-OM) Description: A 34-item self-report questionnaire assessing well-being, problems/symptoms, functioning, and risk. Each item is rated on a 5-point scale (0 = "not at all" to 4 = "most or all of the time"). Higher scores indicate greater distress.

CONTACTS AND LOCATIONS:
Overall Officials: Fabio Leonardi, Psychologist, Principal Investigator — Private Practice, Livorno (Italy)
Locations (2):
- Italy (2):
  - Studio di psicoterapia Dr. Tinacci, Empoli, Italy
  - Studio di Psicoterapia Dr. Fabio Leonardi, Livorno, Li

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be available for five years from the date of the first publication.
Access Criteria: Any researcher can access the data by sending an email to the study coordinator at dott.leonardifabio@gmail.com.

REFERENCES:
- [Background] Strupp, H. H., Horowitz, L. M., & Lambert, M. J. (Eds.). (1997). Measuring patient changes in mood, anxiety, and personality disorders: Toward a core battery. Washington, DC: American Psychological Association.
- [Background] Lyne KJ, Barrett P, Evans C, Barkham M. Dimensions of variation on the CORE-OM. Br J Clin Psychol. 2006 Jun;45(Pt 2):185-203. doi: 10.1348/014466505x39106. PMID 16783905
- [Background] Weiner IB. Psychotherapy relationships that work: therapist contributions and responsiveness to patients. Psychother Res. 2003 Jan 1;13(4):529-32. doi: 10.1093/ptr/kpg044. No abstract available. PMID 21827260
- [Background] Kazi M. (2003). Realist evaluation for practice, British Journal of Social Work, 33, 6, 803-818.
- [Background] Kazdin AE. The meanings and measurement of clinical significance. J Consult Clin Psychol. 1999 Jun;67(3):332-9. doi: 10.1037//0022-006x.67.3.332. PMID 10369053
- [Background] Jacobson, N.S., Follette W.C., Revenstorf D. (1984). Psychotherapy outcome research: methods for reporting variability and evaluating clinical significance, Behaviour Therapy, 15, 336-52.
- [Background] Evans, C., Mellor-Clark, J., Margison, F., Barkham, M., McGrath, G., Connell, J., Audin, K. (2000). Clinical outcomes in routine evaluation : the CORE-OM. Journal of Mental Health, 9, 247-55.
- [Background] Evans, C., Connell, J., Barkham, M., Marshall, C., & Mellor-Clark, J. (2003). Practice-based evidence: Benchmarking NHS primary care counselling services at national and local levels. Clinical Psychology & Psychotherapy, 1, 374-388.
- [Background] Seligman ME. The effectiveness of psychotherapy. The Consumer Reports study. Am Psychol. 1995 Dec;50(12):965-74. doi: 10.1037//0003-066x.50.12.965. PMID 8561380
- [Background] Lambert, M. J. (2004). Ed. Handbook of Psychotherapy and Behavior Change. 5th ed. New York, NY: John Wiley & Sons Inc.
- [Background] Weakland, J. H., Fisch, R., Watzlawick, P., & Bodin, A. (1974). Brief therapy: Focused problem resolution. Family Process, 13, 141-168.
- [Background] Haley, J. (1987). Problem- Solving therapy: New strate- gies for effective family therapy (2nd ed.). San Francisco: Jossey-Bass.
- [Background] Fisch, R., Weakland, J. H., & Segal, L. (1982). The tactics of change: Doing therapy briefly. San Francisco: Jossey-Bass.
- [Background] Rohrbaugh, M. (1986). Q-sort comparisons of the structural, strategic, and systemic family therapies. American Journal of Family Therapy, 14, 40-48.